CLINICAL TRIAL: NCT06445309
Title: Design and Development of a Functional Plant-based Beverage Formulated According to the Main Nutritional Guides for Early Elderly Requirements to Improve Nutritional Status and Immunity for the Early Elderly People to Get Well-healthy Ageing
Acronym: IMMUGOLD
Status: Not yet recruiting | Type: Observational
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Rosa Sola, Clinical professor, University Rovira i Virgili
Other Study IDs: CEIPSA-2023-PR-0024
Record Dates: First submitted 2024-05-15; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Between 80-100 healthy volunteers between 60-75 years old are needed to carry out this sensory tasting study in untrained tasters.
  Additionally, the participant will be given a form to assess the Geriatric Oral Health Assessment Index (GOHAI) and a form for the assessment of dysphagia (EAT-10) to assess the participant's sensory perceptions, as well as any oral health problems. oral health that could interfere with the results of the sensory tasting.
  Interventions: Other: Sensory test of functional plant-based drink

INTERVENTIONS:
Other: Sensory test of functional plant-based drink — Once the volunteers have been recruited, a telephone interview lasting less than 10 minutes will be carried out where what the study consists of will be explained as well as the information sheet for the participant will be read to them so that they understand what the study consists of. study. Once the necessary questions have been asked according to the inclusion criteria, if the participant enters the study, data such as name, surname, age, gender, smoker, consumer of vegetable drinks, pathologies and contact information will be collected. If the participant does not enter the study, their personal data will no longer be collected and they will be informed that according to the exclusion criteria they can no longer participate in the study. Once these data are obtained, it will be randomized using the EXCEL program.

SUMMARY:
Populations around the world are aging and this demographic transition will impact almost every aspect of society. Furthermore, the COVID-19 pandemic has highlighted the seriousness of gaps in policies, systems and services. According to the World Health Organization (WHO) plan for 2021-2030, a decade of concerted global action on healthy ageing is urgently needed to ensure that older people can realize their potential in dignity and equality in nutritional requirements. An effective way to address the inherent demographic change, which translates into the health status of older people, is through the maintenance of adequate nutritional status. Public health services require new funding to address this problem, but if we bring new strategies to health policies, by improving nutrition, we could impact the reduction of costs at the level of medical care in the ageing population. In older people, according to the latest guidelines on nutritional requirements in geriatrics from the Spanish Nutrition Foundation (FEN), the British Nutrition Foundation and The European Society for Clinical Nutrition and Metabolism (ESPEN), multinutrient strategies instead of mononutrient strategies, are gaining importance due to relevant scientific evidence based on controlled and randomized clinical trials. Therefore, following the nutritional requirements in healthy ageing, an important aspect is to strengthen immunity in this population.

Consequently, the food industry is booming in the development of new functional alternatives, such as plant-based beverages, which are well positioned in the market and can offer healthy functional beverage options to people of early elderly age (60 to 75 years) as a target population due to the ease with which they are ingested. Therefore, investments in small and medium-sized companies to encourage the incorporation of trained doctoral personnel and add innovation value to this type of product are essential for resilience.

Therefore, the present proposal hypothesizes that, following the nutritional needs for healthy ageing, a multinutrient-optimized beverage as a functional food can improve immunity and reduce inflammation and oxidation in women and men in the elderly population.

ELIGIBILITY:
Inclusion criteria:

- Men or women ≥60 years old <75 years old; Written informed consent provided prior to the sensory tasting study.

Exclusion Criteria:

* Type 2 diabetes
* Chronic alcoholism
* Early community-dwelling seniors
* Failure to comply with study guidelines.

Selection criteria

Volunteers will be recruited through several ways:

* general databases of participants from previous clinical trials of the NFOC-Salut group
* Leaflets with study information, as well as contact information, will be distributed in health centers, civic centers and social centers.
* The information will be disseminated through brochures with contact information among the people who are registered in the IMSERSO to select those who meet the inclusion criteria according to the study population in order to reach the largest number of subjects possible.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between 80-100 healthy volunteers between 60-75 years old are needed to carry out this sensory tasting study in untrained tasters, the target population of this functional drink. According to Gacula and Rutenbeck, 2005, The sample size ranges from 20 to 200 to detect a difference ranging between 0.0 and 1.0 on a 9-point hedonic scale. For the simulated consumer data, the significant difference was first observed with a difference of 0.60 when n = 40. Factors such as the age of the participants and the number of sensory attributes it is recommended to increase the number of participants, concluding that Between 40-100 participants would be enough to observe a difference above 0.6. Furthermore, according to the European Sensory Network, 2011, for sensory tasting studies with hedonic attributes, between 80-100 participants are recommended.
  All participants will try the same vegetable drink.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Sensory test of a functional plant-based drink | immediatly after intervention
  Sensory attributes will be assessed.

SECONDARY OUTCOMES:
Oral health | immediatly after intervention
  To test the oral health of the early elderly population. Geriatric Oral Health Assessment Index (GOHAI TEST). Consists in a little questionnaire of 12 questions items classified by Yes, always; F, frequently; AV, sometimes; RV, rarely; N, never.
Dysphagia | immediatly after intervention
  To test the dysphagia status of the early elderly population. Eating Assessment Tool EAT-10 TEST. Consists in a little questionnaire of 10 items classified punctued betwen 0-4 being 0 any problem and 4 severe problem.

IPD SHARING:
Plan to Share IPD: No